CLINICAL TRIAL: NCT00976235
Title: Five Year Follow up of IMT-002 Patients; A Long-Term Monitoring Study of IMT-002 Patients
Brief Title: A Long-Term Monitoring Study of the IMT-002 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMT-002-LTM
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Visual Impairment; Quality of Life; Telescope Prosthesis
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMT (Experimental)
  Interventions: Device: IMT - Implantable Miniature Telescope

INTERVENTIONS:
Device: IMT - Implantable Miniature Telescope — Implantation of the telescope prosthesis (performed under the initial study)

SUMMARY:
This is a 5-year study of patients implanted with the Implantable Miniature Telescope (IMT by Dr. Isaac Lipshitz) under Protocol IMT-002. All patients implanted with the telescope prosthesis who enrolled in the IMT-002 trial were asked to participate in this study to monitor long-term safety. Patients will undergo examinations at six-month intervals up to a total of 5 years following implantation.

DETAILED DESCRIPTION:
Every 6 months, manifest refraction, visual acuity, intraocular pressure, slit lamp examination, endothelial cell density, device failures, complications and adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have participated in the IMT-002 trial.
* Patients must be able to understand and comply with the requirements of the clinical study, and be able to abide by the requirements and restrictions of the study.
* Patients must be able to provide voluntary informed consent, and must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Patients who have not participated in the IMT-002 trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2006-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Long term safety (Intraocular pressure, Slit lamp, Endothelial Cell Density, Visual Acuity, Complications, Adverse Events and Device Failures) | 5 years from implantation

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Retina Centers P.C., Tucson, Arizona
  - University of California at Irvine, Irvine, California
  - Altos Eye Physician, Los Altos, California
  - Doheny Retina Institute - University of Southern California, Los Angeles, California
  - Sarasota Retinal Institute, Sarasota, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Kraft Eye Institute, Chicago, Illinois
  - Paducah Retinal Center, Paducah, Kentucky
  - Wilmer Ophthalmological Institute, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - W.K. Kellogg Eye Center, Ann Arbor, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Associated Eye Care, Stillwater, Minnesota
  - Discover Vision Centers, Independence, Missouri
  - Manhattan Eye & Ear, New York, New York
  - Southeast Clinical Research, Charlotte, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Fine, Hoffman & Packer, Eugene, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Vitreoretinal Foundation, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Medical Center Ophthalmology, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin